CLINICAL TRIAL: NCT05283655
Title: Heart Rate Variability in Patients With Irritable Bowel Syndrome Before and After Gut-directed Hypnotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gabriele Moser, Head of psychosomatic Gastroenterology Outpatient Clinic, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 179079
Record Dates: First submitted 2021-08-10; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: pre-post intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): 10 weekly sessions of gut-directed hypnotherapy (behavioral intervention).
  Interventions: Behavioral: Gut-directed hypnotherapy

INTERVENTIONS:
Behavioral: Gut-directed hypnotherapy — hypnotherapy

SUMMARY:
Dysregulation of the brain-gut-axis is believed to underlie symptom generation in irritable bowel syndrome (IBS). The Autonomous Nervous System (ANS) is an important route of brain-gut communication and aberrant ANS functioning, reflected in abnormalities in Heart Rate Variability (HRV) have been described in IBS. Gut-directed hypnotherapy (GHT) leads to symptom reductions in IBS and is supposed to increase parasympathetic regulation. To date, however, the role of therapeutic modulation of the ANS through GHT has been rarely examined. Aim of this pilot study is therefore to assess the impact of GHT on ANS functioning as reflected in heart rate variability. 24h-electrocardiogram before and after 10 sessions of gut-directed hypnotherapy will be administered in groups. Time and Frequency measures of Heart Rate Variability (HRV) will be extracted from 24h-electrocardiogram protocols as indicators of ANS regulation. Validated questionnaires will be utilized to assess IBS symptoms (IBS-SSS) and psychological distress (HADS-D).

DETAILED DESCRIPTION:
Background. The autonomous nervous system (ANS) is a key substrate for the regulation of gastrointestinal homeostasis and plays a substantial role in the pathophysiology of IBS. A convincing amount of evidence indicates a relationship between specific patterns of disturbed sympathovagal balance, symptom severity, and IBS subtypes. According to the literature, hypnosis affects sympathovagal balance by inducing elevated parasympathetic nervous system activity and reduced sympathetic tone. Previous studies reported clinical improvements of IBS-symptoms after successful Gut-directed group Hypnotherapy (GHT) over long-term periods but rarely depicted the underlying alterations in ANS regulation.

Aims of the study. The aim of this study is to investigate short- and long-term effects of Gut- directed group Hypnotherapy (GHT) on ANS regulation in refractory IBS-subjects, measured by heart rate variability. We further attempt to reveal differences in effects of GHT treatment on ANS regulation between IBS-subtypes (constipation-predominant vs. diarrheapredominant) and examine the relationship between self-rated hypnotic depth and parasympathetic activity. Methods. Within a period of 29 months, a sample of N=50 consecutive IBS-patients receive GHT treatment (7-10 weekly sessions) at the Psychosomatic Out-patient Clinic, Division of Gastroenterology and Hepatology, University Hospital of Vienna. Alterations in heart rate variability (HRV) are extracted by Electrocardiogram (ECG) recording in supine (30 min), sitting (10 min) and standing (10 min) position. HRV indices of sympathetic and parasympathetic control are quantified by using measures from time and frequency domains. Assessment of psychological variables is carried out by standardized questionnaires: anxiety, depression, stress, resilience, quality of life and IBS symptom burden.

Methods. Recordings of heart rate and R-R intervals will be conducted continuously for 24 hours. Electrocardiogram (ECG) recordings will be performed within one week before the first and after the last session of hypnosis. Patients will previously informed about the practical requirements for the recordings as well as the role of heart rate variability for health and the presumed associations between Autonomous Nervous System function, psychological stress reactivity patterns and digestive function. Recording devices will be mounted and activated at the hospital. Patients will return to their home or work environment and will be instructed not to ingest stimulating drinks (such as coffee, energy drinks), alcohol and not to engage in physical exercises during the whole recording time. Patients will return to the hospital >24h later for removal and readout of the recording devices. Recorded data will be transferred to Kubios HRV® analysis software (version 2.2, Kuopio, Finland) for subsequent analysis. Calculated parameters comprise mean heart rate, square root of the mean squared differences of successive RR intervals (RMSSD), standard deviation of the normal-to-normal interval (SDNN) in the time domain, and and the number of pairs of succession normal-to-normal intervals that differ by more than 50ms divided by the total number of normal-to-normal intervals (pNN50); in the frequency domain low frequency (0.04-0.15 Hz, LF) and high frequency (0.16-0.40 Hz, HF) will be considered as proposed by international guidelines.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of IBS classified by Rome-IV-criteria
* refractory to diet interventions and symptomatic IBS-medications
* age between 18 and 70 years

Exclusion Criteria:

* pregnancy
* diabetes mellitus
* untreated thyroid disease
* cardiovascular disorders or arrhythmias
* medications possibly interfering with heart rate variability
* nicotine consumption
* bowel surgery
* mental retardation
* current history of severe psychiatric disorder
* over one hour driving time to the hospital

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-12-07 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability | 24 hours
  Standard Deviation of the NN-Interval (SDNN)

SECONDARY OUTCOMES:
Irritable bowel syndrome symptom severity | 10 days
  Irritable bowel syndrome - severity scoring system (IBS-SSS), a questionnaire for clinical assessment of IBS symptom burden and severity. Values range between 0 and 500, with higher values representing higher symptom burden. Values can be classified as mild (values ranging between 75-175), moderate (175-300), and severe (300-500).

IPD SHARING:
Plan to Share IPD: No